CLINICAL TRIAL: NCT05478174
Title: A Multicenter, Randomized, Double-blinded, Propofol-controlled, Phase 3 Clinical Study to Evaluate the Efficacy and Safety of HSK3486 Injectable Emulsion for Induction of General Anesthesia in Adults Undergoing Elective Surgery
Brief Title: Efficacy and Safety of HSK3486 Compared to Propofol for Adults Undergoing Elective Surgery With General Anesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco-USA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSK3486-305
Record Dates: First submitted 2022-07-22; First posted 2022-07-28 (Actual); Results first posted 2024-10-29 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-09

CONDITIONS: General Anesthesia
MeSH Terms: interventions — HSK3486; Propofol

STUDY DESIGN:
Intervention Model Description: Surgical pre-induction analgesia
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded, 2:1 ratio of HSK3486 and Propofol respectively
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HSK3486 (Experimental): HSK3486 for general anesthesia induction
  Interventions: Drug: HSK3486
- Propofol (Active Comparator): Propofol for general anesthesia induction
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: HSK3486 — HSK3486 for induction of general anesthesia
  Arms: HSK3486
Drug: Propofol — Propofol for induction of general anesthesia.
  Other Names: Diprivan
  Arms: Propofol

SUMMARY:
To demonstrate HSK3486 0.4/0.2 mg/kg (0.4 mg/kg intravenous [IV] slow injection over 30 [±5] seconds for the first dose, an additional 0.2 mg/kg if needed) is non-inferior to propofol 2.0/1.0 mg/kg (2.0 mg/kg IV slow injection over 30 [±5] seconds for first dose, an additional 1.0 mg/kg if needed) in success of induction of general anesthesia in adults undergoing elective surgery.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blinded, propofol-controlled, phase 3 clinical study to evaluate the efficacy and safety of HSK3486 for induction of general anesthesia in adults undergoing elective surgery with endotracheal intubation.

After screening, eligible subjects will be randomized in a 2:1 ratio to receive either HSK3486 0.4/0.2 mg/kg (i.e., 0.4 mg/kg IV slow injection over 30 [±5] seconds followed by an additional 0.2 mg/kg dose over 10 [±2] seconds if needed) or propofol 2.0/1.0 mg/kg (i.e., 2.0 mg/kg IV slow injection over 30 [±5] seconds followed by an additional 1.0 mg/kg dose over 10 [±2]seconds if needed) in a blinded manner. Enrolled subjects will be stratified by American Society of Anesthesiologists Physical Status (ASA-PS; I-II and III-IV), age (<65 and ≥65 years), and Body Mass Index (BMI <35 and ≥35 kg/m2). Endotracheal intubation will be performed after adequate anesthetic induction (Modified Observer's Assessment of Awareness/Sedation [MOAA/S] ≤1) (Appendix 1) has been achieved and administration of neuromuscular blocking agent.

Before surgery, premedication is allowed except for sedative-hypnotic or analgesic drugs. Premedication should be recorded if used.

Prior to administration of the study drug in the operating room, the preoperative readiness of each subject will be confirmed. Oxygen will be supplied through a facemask (oxygen flow rate: ≥4 L/min) at least 2 minutes before study drug administration. Subsequently, the investigator can adjust the oxygen flow according to the specific situation of the subject and maintenance IV solution (normal saline [NS], lactated ringer's [LR], or 5% dextrose) will be administrated through IV infusion. Throughout the preinduction and induction periods, a timing device must be used to allow accuracy and sequencing of necessary assessments.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects undergoing elective surgery (non emergency, non cardiothoracic, and non intracranial surgery, anticipated to last at least 1 hour) requiring endotracheal intubation and inhalation general anesthesia during the maintenance period. Duration of surgery is defined as time from study drug administration to time of transfer from operating room to recovery room or PACU.

  2. Males or females, aged ≥18 years old, with ASA-PS I to IV (Appendix 6). For ASA-PS IV subjects, clinical status must be optimized at time of preoperative anesthesia evaluation per judgement of the anesthesiologist.

  3. BMI ≥18 kg/m2. 4. Vital signs at screening: RR ≥10 and ≤24 breaths/min; SpO2≥92% in ambient air; SBP ≥90 and ≤160 mmHg; DBP ≥55 and ≤100 mmHg; HR ≥55 (or ≥50 if subjects are on beta blockers) and ≤100 beats/min.

  5. For all women of childbearing potential, negative serum pregnancy test at screening and must have negative urine pregnancy test at baseline (Day 1). Additionally, women of childbearing potential* must agree to use effective contraception as defined in 7.3.4 from the time of consent until 30 days post study drug administration.

  6. Capable of understanding the procedures and methods of this study, willing to sign an Informed Consent Form, and able to complete this study in strict compliance with the study protocol.

  7. Willing to comply with the site's COVID guidelines and testing requirements as applicable.

  8. Patients with psychiatric/mental disorders must be considered stable on treatment (e.g., SSRIs, SNRIs, TCAs, MAOIs, psychotherapy) and no hospitalizations and urgent care for at least 1 year.

  *Women NOT of childbearing potential are defined as those who have been surgically sterilized (hysterectomy, bilateral salpingo-oophorectomy) or who are postmenopausal (defined 12 months since last regular menses).

Exclusion criteria:

1. Contraindications to deep sedation/general anesthesia or a history of adverse reaction to sedation/general anesthesia.
2. Known to be allergic to eggs, soy products, opioids and their antidotes, or propofol; subject having contraindications to propofol, opioids, and their antidotes.
3. Medical condition or evidence of increased sedation/general anesthesia risk as follows:

   1. Cardiovascular disorders: uncontrolled hypertension (SBP>160 mmHg and/or DBP >100 mmHg) with or without antihypertensive therapy (antihypertensive therapy should be stable for 1 month prior to screening), serious arrhythmia (including the subjects with implanted pace makers), unstable heart failure, Adams-Stokes syndrome (i.e., syncope or near syncope due to cardiac arrythmia), unstable angina, myocardial infarction occurring within 6 months prior to screening, history of tachycardia/bradycardia requiring medications, third degree atrioventricular block or QT interval corrected for HR using Fridericia's formula (QTcF)≥450ms for males and ≥470ms for females.
   2. History of severe obstructive lung disease (i.e., forced expiratory volume in 1 second [FEV1] <50% predicted), history of bronchospasm requiring treatment in a hospital emergency room or hospitalization occurring within 3 months prior to screening, developing acute respiratory tract infection within 2 weeks prior to baseline (such as symptoms of fever, shortness of breath, wheezing, nasal congestion, and cough).
   3. Cerebrovascular disease: subject with a history of serious craniocerebral injury, convulsion, seizure disorder, intracranial hypertension, cerebral aneurysm, or stroke.
   4. Patients with psychiatric diseases (schizophrenia, mania) who have not been on a stable treatment regimen (with SSRIs, SNRIs, TCAs, MAOIs) for at least 1 year or who have been hospitalized or had emergent/urgent care within the past year.
   5. Uncontrolled clinically significant conditions of liver (e.g., severe hepatic insufficiency defined as Childs-Pugh class C), kidney, gastrointestinal tract, blood system, nervous system, or metabolic system diseases, judged by the investigator to be unsuitable for involvement in the study.
   6. Known glycosylated hemoglobin (HbA1c) greater than or equal to 10%.
   7. Known thyroid-stimulating hormone (TSH) value 10% outside the normal range or on thyroid replacement therapy with a known free T-4 level outside the normal range.
   8. History of alcohol abuse within 3 months prior to screening, where alcohol abuse refers to daily alcohol drinking >2 units (1 unit = 360 mL of beer or 45 mL of spirit with a strength of 40% or 150 mL of wine).
   9. History of drug abuse that, in the opinion of the investigator, may confound the interpretation of safety or efficacy in a study subject.
4. Management risks of respiratory tract and judged by the investigator to be unsuitable for inclusion in the study as follows:

   1. Asthma must be stable: stable doses of asthma medications for the past 6 months, no requirement for rescue inhalers or oral steroids within past 6 months, not evaluated in emergency department, urgent care, or hospitalized for an asthma attack within past 1 year.
   2. History (or family history) of malignant hyperthermia.
   3. Any previous failure of tracheal intubation.
   4. Judged to have a difficult airway for endotracheal intubation in the opinion of the Investigator based on parameters such as modified Mallampati score (Grade III or IV [Appendix 7], neck mobility, short thyromental distance, and/or history of difficult intubation).
5. Any medication that has the potential to interact synergistically with propofol or HSK3486, including but not limited to all sedatives and hypnotics (e.g., benzodiazepines and opioids) taken within 5 half-lives prior to Day 1.
6. Laboratory parameters measured at screening with the following levels:

   1. Neutrophil count ≤1.5 x 109/L
   2. Platelet count <80 x 109/L
   3. Hemoglobin <90 g/L (without blood transfusion within 14 days)
   4. Alanine transaminase and/or aspartate transaminase ≥2.0 x upper limit of normal (ULN)
   5. Total bilirubin ≥2.0 x ULN
   6. Severe renal impairment defined by creatinine clearance (CrCl) ≤30 mL/min
7. Female subjects with a positive pregnancy test at screening (serum) or baseline (urine); lactating subjects; any subject planning to get pregnant within 1 month after the study (including the male subject's partner).
8. Judged by the investigator to have any other factors that make the subject unsuitable for participation in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Shoals Medical Trials, Inc., Sheffield, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - UC Davis Health, Davis, California
  - Coastal Clinical Research Specialists, Jacksonville, Florida
  - University of Miami Hospital, Miami, Florida
  - Gulfcoast Research Institute, Llc, Sarasota, Florida
  - Phoenix Clinical Research, Tamarac, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - NextStage Clinical Research - Abay Neuroscience Center, Wichita, Kansas
  - Chesapeake Research Group, Llc, Pasadena, Maryland
  - Brigham & Women'S Hospital, Boston, Massachusetts
  - Duke University Health, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - HD Research, Bellaire, Texas
  - Hd Research Llc., Carrollton, Texas
  - The University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Urology San Antonio Research, San Antonio, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Jbr Clinical Research, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HSK3486 | Propofol
Started | 267 | 133
Dosed | 255 | 129
Full Analysis Set | 255 | 128
Safety Set | 255 | 129
Completed | 254 | 129
Not Completed | 13 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HSK3486 | Propofol | Total
Number analyzed (Participants) | 255 | 128 | 383
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 192 | 97 | 289
  >=65 years | 63 | 31 | 94
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 153 | 84 | 237
  Male | 102 | 44 | 146
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 16 | 50
  Not Hispanic or Latino | 220 | 110 | 330
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 41 | 20 | 61
  White | 203 | 102 | 305
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 2 | 4 | 6
ASA-PS [Count of Participants; unit: Participants] — ASA-PS is evaluated preoperatively at the screening visits per judgement of the anesthesiologist:
  ASA I: Normal and healthy. No systemic diseases other than local lesions. ASA II: A subject with mild systemic disease. ASA III: A subject with severe systemic disease that results in functional limitations but not incapacity. ASA IV: A subject with severe systemic disease that is a constant threat to life and results in incapacity. ASA V: A moribund subject who is not expected to survive without the operation.
  Participants
    ASA-PS I | 62 | 27 | 89
    ASA-PS II | 135 | 74 | 209
    ASA-PS III | 58 | 27 | 85
BMI [Count of Participants; unit: Participants]
  <35kg/m^2 | 204 | 102 | 306
  ≥35kg/m^2 | 51 | 26 | 77

OUTCOME MEASURES:

1. Primary Outcome: Success Rate of General Anesthesia Induction
Description: 1. Induction success (MOAA/S ≤1) after administration of the study drug, and
  2. One or less top-up doses required without using any rescue drugs.
Time Frame: From the time of study drug administration to desired depth of anesthesia to MOAA/S≤1 ( up to 5 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | HSK3486 | Propofol
Number analyzed (Participants) | 255 | 128
Participants | 253 | 128
Statistical Analysis 1: Comparison: HSK3486 vs Propofol; Test type: Non-Inferiority — Non inferiority margin is -8%; p < 0.001, Farrington-Manning method — P-Value for non inferiority test; Risk Difference (RD) = -0.0078, 95% CI 2-sided [-0.0411 to 0.0255]

2. Secondary Outcome: Percentage of Subjects With Successful Induction Who Maintain the Desired Depth of Anesthesia for General Elective Surgery, AND Without Significant Cardiac and Respiratory Depression
Description: The outcome is defined by all the following conditions:
  a) Desired depth of anesthesia for general elective surgery is defined if all following criteria are met: i) No clinical signs of inadequate depth of anesthesia, such as lacrimation, movement, vomiting, coughing, laryngospasm, bucking, swallowing reflex or bronchospasm etc.
  ii) No blood pressure (SBP, DBP, or MAP) increases more than 20% from baseline in response to any major operational procedures or noxious stimulus in defined period.
  iii) Subjects maintain desired depth of anesthesia for general elective surgery with BIS as an objective assessment (after reaching initial lowest value, BIS remains sustainable level at not more than 60).
  b) No significant respiratory depression, such as apnea, prior to the administration of rocuronium bromide.
  c) No significant cardiac depression indicated by blood pressure decrease that requires intervention, i.e., vasopressors and/or IV fluid resuscitation.
Time Frame: 15 minutes from end of drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | HSK3486 | Propofol
Number analyzed (Participants) | 255 | 128
Participants | 88 | 53
Statistical Analysis 1: Comparison: HSK3486 vs Propofol; Test type: Superiority; p = 0.171, Cochran-Mantel-Haenszel; Risk Difference (RD) = -0.0716, 95% CI 2-sided [-0.1742 to 0.0310]

3. Secondary Outcome: Percentage of Subjects With Any Injection-site Pain on Numeric Rating Scale ≥1
Description: 0 = No Pain 1-3 = Mild Pain 4-6 = Moderate Pain 7-9 = Severe Pain 10 = Worst pain imaginable
Time Frame: From start of drug administration to MOAA/S ≤1 (up to 3 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | HSK3486 | Propofol
Number analyzed (Participants) | 255 | 128
Participants | 42 | 58
Statistical Analysis 1: Comparison: HSK3486 vs Propofol; Test type: Superiority; p < 0.001, ANOVA; Mean Difference (Final Values) = -1.76, 95% CI 2-sided [-2.22 to -1.31], Standard Error of Mean 0.231

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) will be collected from the time of informed consent until the final study visit (Day 8). A treatment-emergent AE is defined as: an AE that occurs after the subject starts treatment with the IMP. If an Investigator becomes aware of a serious adverse event within 30 days after the last dose of study drug and it is considered by him/her to be caused by the study drug with a reasonable possibility, the event must be documented and reported.
Description: Adverse Events of Special Interest (AESIs) due to pharmacological effect of an anesthetic agent include hypoxemia, bradycardia, severe hypotension, allergy/anaphylaxis, cardiac arrhythmia and QTc prolongation.
Arm/Group | HSK3486 | Propofol
All-Cause Mortality (participants affected / at risk) | 0/255 | 0/129
Serious Adverse Events (participants affected / at risk) | 6/255 | 2/129
Other Adverse Events (participants affected / at risk) | 178/255 | 89/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HSK3486 (N=255) | Propofol (N=129)
Hypotension (Vascular disorders) | 1 | 0
Post-procedural hemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Ischemic stroke (Vascular disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HSK3486 (N=255) | Propofol (N=129)
Hypotension (Vascular disorders) | 52 | 29
Nausea (Gastrointestinal disorders) | 52 | 25
Procedural Pain (Injury, poisoning and procedural complications) | 38 | 24
Asthenia (General disorders) | 36 | 23
Hypertension (Vascular disorders) | 30 | 15
Procedural Hypotension (Vascular disorders) | 21 | 17
Dizziness (Nervous system disorders) | 15 | 6
Vomitting (Gastrointestinal disorders) | 16 | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 14 | 6
Bradycardia (Cardiac disorders) | 13 | 5
Constipation (Gastrointestinal disorders) | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-02-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT05478174/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT05478174/SAP_001.pdf